CLINICAL TRIAL: NCT05794282
Title: Robotic Total Hip Arthroplasty Anesthesia Management: Retrospective Study
Brief Title: Robotic Total Hip Arthroplasty Anesthesia Management
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Umut Kara, Associate Professor, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Other Study IDs: 2023-65
Record Dates: First submitted 2023-03-20; First posted 2023-04-03 (Actual); Last update posted 2023-04-05 (Actual); Status verified 2023-03

CONDITIONS: Hip Osteoarthritis; Joint Diseases; Anesthesia
MeSH Terms: conditions — Osteoarthritis, Hip; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group rTHA (robotic total hip arthroplasty): the robot assisted total hip arthroplasty
  Interventions: Procedure: the robot assisted total hip arthroplasty
- Group cTHA (conventional total hip arthroplasty): the conventional total hip arthroplasty
  Interventions: Procedure: the conventional total hip arthroplasty

INTERVENTIONS:
Procedure: the robot assisted total hip arthroplasty — the robot assisted total hip arthroplasty
  Groups: Group rTHA (robotic total hip arthroplasty)
Procedure: the conventional total hip arthroplasty — the conventional total hip arthroplasty
  Groups: Group cTHA (conventional total hip arthroplasty)

SUMMARY:
Robotic arthroplasty is increasing in acceptance on a global scale as a result of advancements in orthopedic surgery technology. The investigators aimed to share their anesthesia management experience as well as compare robotic unilateral total hip arthroplasty with conventional surgical technique in this retrospective study.

DETAILED DESCRIPTION:
This study was conducted after obtaining ethics committee approval.

The inclusion criteria were as follows: American Society of Anesthesiologists (ASA) physical status I-III patients between 40-85 years, elective unilateral THAs which were performed by a single senior orthopedic surgeon and orthopedic team between January 2021 and January 2023 under CSEA. Exclusion criteria were urgent surgery, bilateral surgery, previous surgery, missing data, and lost to follow-up in the perioperative period.

The routine anesthetic protocol for the TKA was as follows: A single dose of 0.5% hyperbaric bupivacaine between 15-10 mg was administered intratechally. Following this the epidural catheter was inserted 4 cm into the epidural space through the epidural needle and secured. The level of the sensory block was assessed using pin-prick and cold sensation tests, and motor block using the Bromage scale. The patients were followed in the postanesthesia care unit (PACU) after the surgery. Patients with a modified Aldrete scoring system ≥9 were considered to be eligible for the transfer from PACU to the service.

Pain was evaluated using a Visual Analogue Scale (VAS) with regular intervals. Data were collected from hospital's electronic database records, patient files, and anesthesia charts.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status I-III
* Between 40-85 years
* Elective unilateral THAs which were performed by a single senior orthopedic surgeon
* Between January 2021 and January 2023 under CSEA.

Exclusion Criteria:

* Urgent surgery
* Bilateral surgery
* Previous surgery
* Missing data and lost to follow-up in the perioperative period

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with American Society of Anesthesiologists (ASA) physical status I-III and elective unilateral THAs between the ages of 40 and 85 will be analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Time | Only in surgery time, an average of 3 hours]
  The duration of surgical procedures

SECONDARY OUTCOMES:
Complications | After the end of surgery, in the first 1-month follow-up
  Perioperative complications rates
Hospital discharge time | Time from discharge from PACU to discharge from hospital, an average of 96 hours
  Time from the beginning of the operation to the discharge of hospital

IPD SHARING:
Plan to Share IPD: Undecided